CLINICAL TRIAL: NCT02089048
Title: An Open Label, Multiple Dose Study to Evaluate the Pharmacokinetics of Auranofin Following Oral Dose Administration for 7 Days to Healthy Subjects
Brief Title: Auranofin PK Following Oral Dose Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-0101; HHSN272200800024C
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2014-03-12

CONDITIONS: Amoebiasis
Keywords: Amebiasis; auranofin; pharmacodynamics; pharmokinetics
MeSH Terms: conditions — Amebiasis | interventions — Auranofin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cohort 1 (Experimental): 15 subjects receive 6mg of auranofin once every 24 hours for 7 days
  Interventions: Drug: Auranofin

INTERVENTIONS:
Drug: Auranofin — Auranofin is a gold-containing chemical salt available as 3mg capsules. Cohort 1 receives 6mg oral dose of auranofin once every 24 hours for 7 days

SUMMARY:
Phase I, open-label study in 15 healthy adult subjects receive 6 mg of auranofin orally once every 24 hours for 7days. Blood samples will be taken for 17 weeks following the last dose of auranofin for determination of terminal phase pharmacokinetic parameters. Stool samples will also be obtained for the measurement of gold.

DETAILED DESCRIPTION:
Auranofin is a gold-containing chemical salt, granted as an orphan drug status for use in the treatment of amebiasis. Amebiasis is a parasitic infection caused by the protozoon Entamoeba histolytica. It affects about ten percent of the world's population, being especially common in areas with poor health infrastructure. This is a Phase I open label, multiple dose study to evaluate the pharmacokinetics of Auranofin following oral dose administration for 7 days to healthy subjects. 15 healthy male and female volunteers age 18-45 years, inclusive enrolled in one site. The study duration is 48 weeks and up to 23 weeks of subject participation. The primary objective characterizes the pharmacokinetics of gold, given as auranofin, during and after 7 days of once daily oral dose administration. The secondary objective monitor the safety of Auranofin during and after 7 days of oral administration.

ELIGIBILITY:
Inclusion Criteria:

-Personally signed and dated informed consent document. -Healthy male or female of non-childbearing potential, between the ages of 18 and 45 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, complete physical examination including vital signs, and clinical laboratory tests. Non-childbearing potential is defined as amenorrheic for at least 2 years plus a serum follicle-stimulating hormone (FSH) level > 30 IU/L, or documented bilateral oophorectomy and/or hysterectomy, or tubal ligation. -Body mass index (BMI) of 18 to 30 [weight (kg)]/ [height (m)^2] inclusive; and a total body weight > 50 kg (110 lbs) and < 122 kg (250 lbs) at the Screening Visit. -Male subjects willing to use appropriate contraception for the duration of the study. -Willing and able to comply with scheduled visits, dosing plan, laboratory tests, and other study procedures.

Exclusion Criteria:

-Evidence or history of clinically significant hematologic, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, musculoskeletal, immunologic, neurologic or dermatologic disease (including drug allergies that are clinically significant) which in the opinion of the Investigator could impact the participation of the subject in the study or the assessment of the study endpoints. -Current evidence of or history of malignancy (excepting completely treated cervical cancer in situ or intraductal carcinoma of the breast, or </= 2 basal cell and/or squamous cell carcinomas of the skin completely excised) in the 5 years prior to Day -1 with no evidence of recurrence. -Breastfeeding or a positive serum pregnancy test at the Screening Visit or Day -1. -History of drug abuse within 6 months prior to study drug administration. -A history of alcohol abuse, defined as regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for men (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor), within 6 months prior to study drug administration. -Positive results from a standard urine drug screen (Screening Visit or Day -1) or a positive test for alcohol (Screening visit or Day -1). -Daily use of tobacco- or nicotine-containing products (cigarettes, pipe, cigar, chewing tobacco or nicotine gum, lozenges or patches). Occasional social smoking is acceptable. You must not change your use of tobacco from your first visit and through completion of the last visit of the study. -Treatment with an investigational drug within 30 days prior to study drug administration. -Prior exposure to gold-containing products. -Use of any prescription or nonprescription drugs, vitamins, or dietary or herbal supplements within 14 days prior to study drug administration. As exceptions, acetaminophen may be used at doses of </=1 g/day until 24 hours prior to study drug administration. -Blood donation of >/= 1 pint (473 mL) within 30 days prior to study drug administration. -Plasma and platelet donation within 14 days prior to study drug administration. -Screening liver function tests (alanine aminotransferase [ALT] or aspartate aminotransferase [AST]) greater than upper limit of normal (ULN). -Evidence of hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection upon serological testing at the Screening Visit. -Evidence of active infection or febrile illness (e.g., bronchopulmonary, urinary or gastrointestinal) within 7 days prior to study drug administration. -History of allergy to auranofin or any of the excipients in the capsules. (excipients per the package insert of auranofin are listed in Section 6.1) -Any other condition that, in the opinion of the investigator, poses a risk to the safety of the individual or the valid conduct of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-04-02 (Actual); Primary Completion 2014-09-09 (Actual); Study Completion 2015-05-13 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of gold following 7 once daily doses of auranofin | Up to Day 126

SECONDARY OUTCOMES:
Type, frequency and severity of Serious AEs (SAEs) to the end of study | Up to Day 126
Type, frequency and severity of treatment-emergent adverse events (TEAEs) to 14 days after administration of the first dose | 14 Days after first dose

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles Phase I Services - Overland Park, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Capparelli EV, Bricker-Ford R, Rogers MJ, McKerrow JH, Reed SL. Phase I Clinical Trial Results of Auranofin, a Novel Antiparasitic Agent. Antimicrob Agents Chemother. 2016 Dec 27;61(1):e01947-16. doi: 10.1128/AAC.01947-16. Print 2017 Jan. PMID 27821451